CLINICAL TRIAL: NCT06584955
Title: Feasibility of the Use of Weighted Blankets to Improve Sleep Among Patients With Hematological Malignancies
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Gabrielles Angel FDN for Cancer Research (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-0464; NCI-2024-07498 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2024-09-03; First posted 2024-09-05 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Hematological Malignancies
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients more than 200 pounds (Experimental)
  Interventions: Other: Weighted Blanket
- Patients between 150-200 pounds (Experimental)
  Interventions: Other: Weighted Blanket

INTERVENTIONS:
Other: Weighted Blanket — Participants will be given a weighted blanket

SUMMARY:
The goal of this clinical research study is to learn about the effects of weighted blankets on sleep quality in patients with blood cancers. Weighted blankets are heavier blankets that contain inner weight beads. The deep pressure stimulation induced by these blankets can have a calming effect.

DETAILED DESCRIPTION:
Primary Objective:

To determine the feasibility of using weighted blankets to improve Sleep Disturbances (SD) for patients with hematological malignancies in an outpatient setting.

Secondary Objectives:

To explore if weighted blanket use improves sleep as assessed by the ESAS sleep question. A positive response is defined by at least a one-point reduction in ESAS sleep between baseline and day 7 +/-2 days.

To explore if weighted blanket use during a 14-day period improves Insomnia Severity Index (ISI) score.

To explore the response rate in anxiety, where response is defined as a minimum of one-point change in the ESAS anxiety score, between baseline and day 7 +/-2 days after the use of weighted blankets.

To explore if patients are satisfied with the use of weighted blankets as determined by a positive response to at least 2 of the 5 patient satisfaction questions.

To assess safety using NCI CTCAE v5

ELIGIBILITY:
Inclusion Criteria:

1. Outpatient at MD Anderson Cancer Center
2. Adult patients ≥ 18 years
3. Diagnosis of hematological malignancy
4. ESAS Sleep>/=4
5. Performance status as measured by Eastern Cooperative Oncology Practice group (ECOG) score of 2 or below

Exclusion Criteria:

1. Platelet count of 25 or below
2. History of seizures/intracranial metastasis/ sleep apnea/restless leg syndrome/paralysis
3. Weight less than 150 lbs.
4. Attending physician assessment of prognosis with expected life expectancy of <1 month
5. Patients who are unable to tolerate their blankets/sheets in the night due to medical conditions such as pain, peripheral neuropathy, night sweats, hot flashes etc.
6. Patients with difficulty breathing, disorders of poor circulation, fragile skin, rash, or open wounds, or by those who are claustrophobic or cleithrophobic.
7. Prior use of weighted blankets within the past 1-year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Santhosshi Narayanan, MBBS, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org